CLINICAL TRIAL: NCT02420730
Title: Safety, Tolerability and Systemic Pharmacokinetics of AGN-232411 in Healthy Participants and Participants With Dry Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 232411-001
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1A: AGN-232411 Dose A (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose A administered in the study eye once daily for one day, followed by twice daily for 16 days in healthy participants.
  Interventions: Drug: AGN-232411
- Cohort 1B: AGN-232411 Dose B (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose B administered in the study eye once daily for one day, followed by twice daily for 16 days in healthy participants if the safety and tolerability of Dose A in Cohort 1A is acceptable.
  Interventions: Drug: AGN-232411
- Cohort 1C: AGN-232411 Dose C (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose C administered in the study eye once daily for one day, followed by twice daily for 16 days in healthy participants if the safety and tolerability of Dose B in Cohort 1B is acceptable.
  Interventions: Drug: AGN-232411
- Cohort 1: AGN-232411 Vehicle (Placebo Comparator): One drop of Vehicle for AGN-232411 topical ophthalmic solution administered in the study eye once daily for one day, followed by twice daily for 16 days in healthy participants.
  Interventions: Drug: AGN-232411 Vehicle
- Cohort 2A: AGN-232411 Dose A (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose A administered in the study eye once daily for one day, followed by twice daily for 27 days in participants with dry eye disease.
  Interventions: Drug: AGN-232411
- Cohort 2B: AGN-232411 Dose B (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose B administered in the study eye once daily for one day, followed by twice daily for 27 days in participants with dry eye disease if the safety and tolerability of Dose A in Cohort 2A is acceptable.
  Interventions: Drug: AGN-232411
- Cohort 2C: AGN-232411 Dose C (Experimental): One drop of AGN-232411 topical ophthalmic solution Dose C administered in the study eye once daily for one day, followed by twice daily for 27 days in participants with dry eye disease if the safety and tolerability of Dose B in Cohort 2B is acceptable.
  Interventions: Drug: AGN-232411
- Cohort 2: AGN-232411 Vehicle (Placebo Comparator): One drop of Vehicle for AGN-232411 topical ophthalmic solution administered to the study eye once daily for one day, followed by twice daily for 27 days in participants with dry eye disease.
  Interventions: Drug: AGN-232411 Vehicle

INTERVENTIONS:
Drug: AGN-232411 — AGN-232411 topical ophthalmic solution
  Arms: Cohort 1A: AGN-232411 Dose A; Cohort 1B: AGN-232411 Dose B; Cohort 1C: AGN-232411 Dose C; Cohort 2A: AGN-232411 Dose A; Cohort 2B: AGN-232411 Dose B; Cohort 2C: AGN-232411 Dose C
Drug: AGN-232411 Vehicle — Vehicle for AGN-232411 topical ophthalmic solution.
  Arms: Cohort 1: AGN-232411 Vehicle; Cohort 2: AGN-232411 Vehicle

SUMMARY:
This study will examine the safety, tolerability, and systemic pharmacokinetics of up to 3 different concentrations of AGN-232411 topical ophthalmic solution in healthy participants and participants with dry eye.

ELIGIBILITY:
Inclusion criteria:

Stage 1

-Healthy participants.

Stage 2 -Participants with the symptoms of dry eye disease.

Exclusion criteria:

Stage 1

-Known allergies or sensitivities to study medications, fluorescein, or lissamine green

Stage 2

* Known allergies or sensitivities to study medications, fluorescein, or lissamine green
* Allergic ocular disease, ocular trauma, corneal erosions or ulcers, or uveitis within the previous 12 months
* History of any ocular surgery within the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- United States (3):
  - Sall Research Center, Artesia, California
  - Lugene Eye Institute, Glendale, California
  - Montebello Medical Center, Inc., Montebello, California